CLINICAL TRIAL: NCT00339027
Title: HealthSpark: Health Access for Children in Federally-Subsidized Child Care
Status: Completed | Type: Observational
Sponsor: University of Miami (Other)
Collaborators: Health Foundation of South Florida (Other); Ounce of Prevention Fund (Other); The Early Childhood Initiative Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 20040116
Record Dates: First submitted 2006-06-16; First posted 2006-06-20 (Estimated); Last update posted 2021-08-11 (Actual); Status verified 2021-08

CONDITIONS: Asthma; Obesity; ADHD
Keywords: child care centers; community based research; behavioral health; health literacy; unmet healthcare needs
MeSH Terms: conditions — Asthma; Obesity; Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Preschool children: Children aged 3-5 years who are enrolled in federally-subsidized early care and education centers in underserved communities in Miami-Dade County

SUMMARY:
HealthSpark is a community-based research network of childcare centers designed to improve the health of children in Miami-Dade County. HealthSpark is the health component of SPARK (Supporting Partnerships to Assure Ready Kids), a community coalition led by the Early Childhood Initiative Foundation to improve school readiness in Allapattah/Model City and Homestead/Florida City, two underserved Miami-Dade County communities. The goal of HealthSpark I is to identify the health and healthcare needs of preschool children, then help translate evidence-based intervention into community programs.

DETAILED DESCRIPTION:
Preschool children are at risk for developing health problems that affect school readiness and that lead to significant health conditions through adulthood. Several decades of research have demonstrated that early identification and intervention is the best approach to ensuring healthy, successful children and adults. Despite advancements in our understanding of child health, large gaps in services continue; especially for children in poverty and for ethnic/racial minorities. National data supports the persistence of health disparities among children.

In May 2004, the HealthSpark team began to collect data from the parents, child care center directors, and local pediatricians in the two targeted communities. The HealthSpark I sample included 681 assessments of parents with children ages three or four years old, 53 child care center directors, and 30 primary care pediatricians. The parent assessments were conducted in person at the child care center. Additionally, in September 2004 four focus groups were conducted in the three primary languages of the communities, English, Spanish, and Creole. A content analysis was done on these sessions to determine the most prominent issues in each location.

Prevalence rates for obesity (38.0%) and asthma (29.3%) among the children the team surveyed were well above the national averages (20% and 7.4%). Despite high rates of health problems, roughly 10% of families reported not being able to get medical care for their child when they needed it, compared to the national average of 1.7% and a state of Florida average of 3.0%. HealthSpark also discovered that 20.9% of children are not properly restrained in motor vehicles. This statistic raises particularly high concern due to the fact that motor vehicle accidents are a leading cause of death among children and proper restraint in a vehicle is one step towards overcoming this statistic.

Access to health care is especially important for children with special health care needs. Of the total population, 8.7% need or use more medical care, mental health, or educational services than the average child. While this is low in comparison to the national average (12.8%), it still accounts for a significant portion of the population and demonstrates the need to ensure all children have appropriate access to care. Even though the majority of the children HealthSpark surveyed had some form of health insurance, 11.3% did not have any. This number is higher than the national average (9.5%) and raises concern over why specific barriers to access healthcare have not been broken down. During focus group sessions, parents described what specific issues were preventing them from either accessing medical care or not getting their children enrolled in the proper insurance program; these problems varied by region. Families located in the Allapattah/Model City region have access to Jackson Memorial Hospital and clinics but described long waiting times before they were able to see a physician. In contrast, families in Homestead/Florida City had more prevalence of uninsured children and are limited by their lack of access to transportation. Few families have cars and many described having to walk several miles in order to use public transportation. Many parents are not satisfied with the quality of healthcare their children are receiving, especially for families in the Homestead/Florida City area. Among the 43 healthcare professionals who deliver most of the pediatric primary care in these communities, 42.9% are not board-certified and only 26.2% are members of the American Academy of Pediatrics.

In HealthSpark I, we discovered child health issues existed in large part because of the lack of care and resources families in Miami-Dade County are receiving. However, even if every family had access to a high quality pediatrician the health of children in these two areas would not immediately improve. Interventions with a high level of collaboration among child care centers, pediatricians, and health educators will be the first step to improving the health of children within these two communities. In HealthSpark II, the intent is to demonstrate that improved coordination and cooperation among professionals and families will improve child health. The resources already exist in each community. In the initial HealthSpark survey, a network of child care centers and pediatricians interested in improving the health environment of the children in their community were identified. The HealthSpark team plans on helping these professionals come together and form a relationship that will improve and address the health needs of families.

ELIGIBILITY:
Inclusion Criteria:

* Children ages 3 - 5 years, enrolled in one of the designated SPARK child care centers

Exclusion Criteria:

* Children under the age of 3 years or over the age of 5 years
* Children whose parents do not want to participate
* Children whose child care centers do not want to participate

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children aged 3-5 years who are enrolled in federally-subsidized early care and education centers in underserved communities in Miami-Dade County
Sampling Method: Non-Probability Sample
Enrollment: 960 (Estimated)
Dates: Start 2004-05; Primary Completion 2005-03 (Actual); Study Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
Health concerns of parents | Cross-sectional
  Descriptive survey

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey P Brosco, MD, PhD, Principal Investigator — University of Miami
Locations (1):
- University of Miami Mailman Center for Child Development, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No